CLINICAL TRIAL: NCT03034694
Title: The Effect of Dermatology and Teledermatology Consultations on Length of Hospital Admission, 30 Day Readmission Rate, and Antibiotic Use in Patients Presenting With Cellulitis vs Pseudocellulitis in an Academic Inpatient Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Benjamin Kaffenberger, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2015H0393
Record Dates: First submitted 2016-06-04; First posted 2017-01-27 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Cellulitis
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Intervention Model Description: Routine Care vs The use of teledermatology
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine Care (Placebo Comparator): The first group will be randomized to routine care of receiving or not receiving a dermatology consult in the hospitalized setting based on the clinical decision of the hospitalist. The patients will see the research coordinator who will take images and for a teledermatology assessment, however, these assessments will not be placed in the chart and the treating hospitalist will not know.
  Interventions: Other: Routine Care
- Teledermatology INtervention (Experimental): The second arm will be patient randomized to teledermatology intervention. These patients will be imaged by the research coordinator, then the assessment will be placed in the chart for the hospitalist to see although final treatment decisions are still made by the hospitalist.
  Interventions: Other: teledermatology consult

INTERVENTIONS:
Other: teledermatology consult — teledermatology consult
  Arms: Teledermatology INtervention
Other: Routine Care — The patient will undergo imaging but this report will not be put into the chart.
  Arms: Routine Care

SUMMARY:
The effect of teledermatology on length of hospital admission, length of stay, 30 day readmission rate, and antibiotic use in patients presenting with cellulitis vs pseudocellulitis in an academic emergency department setting.

ELIGIBILITY:
Inclusion Criteria:

* Over 18
* Admission for cellulitis-like symptoms, including but not limited to the following: tenderness, redness, swelling, expansive lesion

Exclusion Criteria:

* pregnant
* prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Length of Hospitalization | 60 Days

SECONDARY OUTCOMES:
Readmission rate | 30 Days
Frequency/Use of antibiotics | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin H Kaffenberger, MD, Principal Investigator — OSU Dermatology
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes